CLINICAL TRIAL: NCT06257680
Title: A Single-armed, Open, Phase I Study of ReT01 ACT Injection in the Treatment of Patients With Advanced Solid Tumors
Brief Title: A Phase I Study on ReT01 ACT for the Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aeonvital Biomedicine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ReT221101
Record Dates: First submitted 2024-01-25; First posted 2024-02-14 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ReT01 ACT (Experimental)
  Interventions: Biological: ReT01 ACT

INTERVENTIONS:
Biological: ReT01 ACT — Patients were infused with ReT01 ACT injection after pretreatment, and subjects were closely observed for 24 hours after each infusion.

SUMMARY:
This single-armed, open, phase I study was designed to evaluate the safety and tolerance of ReT01 ACT injection in the treatment of advanced solid tumors. The phase I clinical trial is expected to be finished in 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. They voluntarily signed the informed consent form (ICF) and completed the study procedure and follow-up examination and treatment.
2. Age from 18 to 75 years old, regardless of gender;
3. The ECOG performance status score was 0-1.
4. Advanced solid tumors positive for PAN-CK, confirmed histopathologically or cytologically: Advanced solid tumors that have failed previous standard therapy (disease progression or intolerance), currently have no standard treatment options, or are unable to receive current standard treatment for other reasons Included, but not limited to, driver gene negative non-small cell lung cancer (NSCLC) (except neuroendocrine tumors or mixed types containing >10% of neuroendocrine tumors), primary or metastatic breast cancer (TNBC), and histopathologically or cytologically confirmed patients with at least one prior platinum-based chemotherapy regimen and no more than three prior systemic treatment failures (disease progression or intolerance) Toxicity) of recurrent/metastatic cervical cancer (cervical squamous, adenosquamous, and adenocarcinoma subjects), ovarian cancer, liver cancer, head and neck cancer, and colorectal cancer (CRC);
5. Subjects had at least one eligible tumor lesion/tissue for preparation of ReT01 ACT injection. Fresh cancerous tissue (proximal metastatic lymph node or tumor margin tissue) with a total tumor volume of at least 0.125 cm3 was obtained by conventional surgical or interventional methods. The number of re-TILs in tumor tissue that met the needs of reinfusion and detection was sufficient.
6. The predicted survival time was ≥3 months.
7. After tumor lesion/tissue sampling, the subject still had at least one measurable tumor lesion according to Response Evaluation criteria in Solid Tumors, version 1.1 (RECIST 1.1) criteria.
8. Patients with good organ function (no platelet or cell stimulating factor transfusion within 14 days before enrollment) and laboratory results meeting the following criteria: 1) absolute neutrophil count (ANC) ≥1.0×109/L; 2) platelet count (PLT) ≥80×109/L; 3) hemoglobin (Hb) ≥80 g/L; 4) Serum bilirubin (TBIL) ≤1.5× upper limit of normal (ULN), if the subject has Gilbert's syndrome or liver metastasis TBIL≤3×ULN; 5) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; If liver metastasis existed, ALT and AST≤5×ULN; 6) international normalized ratio (INR) ≤1.5×ULN, activated partial thromboplastin time (APTT) ≤1.5×ULN (except those on anticoagulant therapy); 7) creatinine clearance ≥60 mL/min (calculated by Cockcroft-Gault formula);
9. Toxic effects from previous therapy had resolved to grade 1 or less before enrollment (with the exception of grade 2 or less neurotoxicity from alopecia and chemotherapeutic agents).
10. Women of childbearing age who had a negative blood pregnancy test within 7 days before enrollment; Any male and female patient of childbearing potential must agree to use effective contraception for at least 6 months from enrollment until infusion of the ReT01 ACT injection. According to the investigator's judgment, a patient was considered to be fertile if the patient was biologically capable of having children and had a normal sexual life. Infertile women were required to meet at least one of the following criteria: 1) prior hysterectomy or bilateral oophorectomy, 2) medically confirmed ovarian failure, 3) medically confirmed, physiologic cessation of menstruation for at least 12 consecutive months (excluding use of chemoradiotherapy or estrogen/progestin-based drugs or other pathological factors);
11. The trial protocol was approved and adhered to, as judged by the investigators.

Exclusion Criteria:

1. There were only bone metastases.
2. Central nervous system metastases were present.
3. He had received other previous adoptive cell therapies.
4. Patients received any systemic anti-tumor therapy (including chemotherapy, radiotherapy, molecular targeted therapy, etc.) within 3 weeks before conditioning.
5. Chinese/herbal medicine with anti-tumor indications was received within 1 week before pretreatment.
6. Treatment with prednisone at a dose of 10 mg or more per day or its equivalent systemic corticosteroids (except for inhaled, topical, or physiological replacement therapy) or other immunosuppressive medications within 2 weeks before conditioning.
7. Any major surgery within 4 weeks before screening that was considered by the investigator to be unsuitable for enrollment or any other planned major surgery during the study (excluding the planned surgery for the preparation of Re-TIL cells as specified in the protocol) (The definition of major surgery was based on the grade 3 and 4 procedures specified in the Administrative Measures for the Clinical Application of Medical Technology implemented on May 1, 2009). ;
8. Patients with other malignant tumors within 5 years before screening or at the same time (patients with locally treated malignant tumors that did not require treatment for more than 1 year and had no significant risk of recurrence according to the investigator's judgment were excluded, including but not limited to non-melanoma skin cancer, bladder cancer, etc.);
9. A history of active or suspected autoimmune or inflammatory disease;
10. Previous history of organ transplantation or hematopoietic stem cell transplantation;
11. Presence of any of the following infections: 1) active hepatitis B (hepatitis B surface antigen [HbsAg] positive and hepatitis B virus DNA [HBV-DNA] > 1000 copies /ml); 2) active hepatitis C (positive for hepatitis C virus (HCV) antibody and HCV RNA (HCV-RNA) test > the lower limit of study detection); 3) active systemic infections requiring antibiotics (e.g., sepsis, bacteremia, fungemia, etc.); 4) congenital or acquired immunodeficiency (including but not limited to severe combined immunodeficiency disease, human immunodeficiency virus (HIV) infection, etc.);
12. Vaccination with a live or attenuated vaccine within 4 weeks before conditioning;
13. Patients with severe cardio-cerebrovascular disease including but not limited to: 1) hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg) that is poorly controlled with medical therapy; 2) previous history of hypertensive crisis or hypertensive encephalopathy; 3) cardiovascular and cerebrovascular events, transient ischemic attack, myocardial infarction, unstable angina, and significant vascular disease (including but not limited to aortic aneurysm or proximal arterial thrombosis requiring surgical repair) within 6 months before enrollment; 4) New York Heart Association (NYHA) class ≥II heart failure with left ventricular ejection fraction (LVEF) <50%; Severe arrhythmias uncontrolled by medication (including QTc interval ≥450 ms in men or ≥470 ms in women, calculated according to Fridericia's formula), ongoing or planned use of medications that may prolong the QT interval, or congenital long QT syndrome;
14. Severe respiratory disease (previous or combined history of severe interstitial lung disease, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, or symptomatic bronchospasm); Forced expiratory volume in 1 second (FEV1) <2 L, carbon monoxide diffusion capacity (DLCO) (calibrated) <40%;
15. A clear previous history of a neurological or psychiatric disorder, including epilepsy or dementia;
16. A history of severe allergic reactions to drugs used during the study (including but not limited to cyclophosphamide, fludarabine, IL-2, components of ReT01 ACT injection, gentamicin, etc.);
17. Other conditions considered by the investigator to be inappropriate for participation in the trial (e.g., grade 3 or higher adverse effects from previous immunotherapy).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-02-18 (Estimated); Study Completion 2027-02-18 (Estimated)

PRIMARY OUTCOMES:
Maximal Tolerance Dose | Up to Day 28
Dose Limiting Toxicity | Up to Day 28
Adverse events (AE) | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Assess for Pharmacokinetics (PK) | through study completion, an average of 1 year
  Evaluate the efficacy of ReT01 ACT based on PK which is analyzed by detection data.
Assess for Pharmacodynamics (PD) | through study completion, an average of 1 year
  Evaluate the efficacy of ReT01 ACT based on PD which is analyzed by detection data.
Objective Response Rate (ORR) | through study completion, an average of 1 year
  Evaluate the efficacy of ReT01 ACT based on ORR which is assess by RECIST v1.1.
Progression Free Survival (PFS) | through study completion, an average of 1 year
  Evaluate the efficacy of ReT01 ACT based on PFS which is assess by RECIST v1.1.
Duration of Response (DOR) | through study completion, an average of 1 year
  Evaluate the efficacy of ReT01 ACT based on DOR which is assess by RECIST v1.1.
Disease Control Rate (DCR) | through study completion, an average of 1 year
  Evaluate the efficacy of ReT01 ACT based on DCR which is assess by RECIST v1.1.
Overall Survival (OS) | through study completion, an average of 1 year
  Evaluate the efficacy of ReT01 ACT based on OS which is assess by RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China